CLINICAL TRIAL: NCT01974713
Title: CAN-AIM to PREVENT: CANadian Study, Assessing Inflammatory Markers to PRedict EVents in Nephrology sTudy
Brief Title: Inflammatory Markers and Adverse Outcomes in Chronic Kidney Disease
Acronym: AIMtoPREVENT
Status: Completed | Type: Observational
Sponsor: Institute of Kidney Lifescience Technologies (Other)
Responsible Party: Sponsor
Other Study IDs: 042010
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Chronic Kidney Disease
Keywords: CKD progression; Inflammation; FGF23; Genetic biomarkers
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Longitudinal cohort of patients with chronic kidney disease followed in 3 kidney centers in Ontario. The goal is to determine whether and how rates of renal disease progression are affected by inflammatory markers, FGF23 levels, and genetic polymorphisms

DETAILED DESCRIPTION:
This longitudinal cohort study will follow 2500 prevalent Chronic Kidney Disease (CKD)patients under the care of a nephrologist at 3 Southern Ontario Nephrology centres and all affiliated satellite centres with an estimated Glomerular Filtration Rate (eGFR) less than 60 ml/min to determine the rate of their renal disease progression over a 36 months. All CKD patients older than 18 years of age may be included in this study. This study will analyze, with 6 month serial measurements, conventional biochemical, hormonal and metabolic parameters in addition to the demographics, clinical status, medications and blood and urine samples of these patients. This study will assess the influence of inflammation on FGF23 and genetic polymorphisms that may reflect the processes involved with disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to a nephrologist for evaluation of CKD or those currently seen by a nephrologist, with eGFR less than 60 ml/min
* Patients that are erythropoietin treatment naive
* Transplant patients with failing grafts requiring nephrologists follow-up
* Patients currently not receiving RRT consenting to be in the study
* Adults 18 years of age and older

Exclusion Criteria:

* Functioning Organ transplant
* Life expectancy less than 12 months
* Patients currently receiving RRT or who will likely initiate RRT within 6 months
* Patients unable or contraindicated to receive EPREX® as erythropoietin replacement therapy for the correction of anemia related to CKD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in chronic kidney disease clinic setting
Sampling Method: Non-Probability Sample
Enrollment: 2530 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Renal function at study censure | 3 years
  Estimated glomerular filtration rate after 3 years of follow-up in the study

SECONDARY OUTCOMES:
Dialysis-dependent renal failure | 3 years
  Development of dialysis-dependent renal failure during observation period

CONTACTS AND LOCATIONS:
Overall Officials: Paul Y Tam, MD, Principal Investigator — Kidney Life Science Institute

IPD SHARING:
Plan to Share IPD: Undecided